CLINICAL TRIAL: NCT05381194
Title: The 6-month BPaL(M) Regimen for the Treatment of Patients With MDR/RR-TB: Multicenter, Single-arm, Operational Research, Clinical Trial
Brief Title: BPaL(M) Regimen for the Treatment of MDR/RR-TB
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Pusan National University Hospital (Other); Samsung Medical Center (Other); Seoul National University Hospital (Other); Severance Hospital (Other); Chonnam National University Hospital (Other); The Catholic University of Korea (Other); Chungbuk National University Hospital (Other); Ulsan University Hospital (Other); Soon Chun Hyang University (Other); Incheon St.Mary's Hospital (Other); DongGuk University (Other); National Medical Center, Seoul (Other)
Responsible Party: Principal Investigator, Tae Sun Shim, Clinical professor, MD, PhD, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BPaL(M)
Record Dates: First submitted 2022-05-08; First posted 2022-05-19 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Multidrug- and Rifampicin-resistant Tuberculosis
MeSH Terms: interventions — Clinical Protocols

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- single arm (investigational arm) (Experimental): BPaLM
  Interventions: Drug: BPaL(M) regimen

INTERVENTIONS:
Drug: BPaL(M) regimen — Patients diagnosed with MDR/RR-TB are initially assigned to the BPaLM regimen as a single-arm for treatment initiation. Afterward, if MDR/RR-TB is confirmed to be fluoroquinolone-resistant by molecular or phenotypic DST, the treatment is switched to the BPaL regimen (for 24 weeks). On the other hand, if MDR/RR-TB is confirmed to be fluoroquinolone-susceptible, treatment for MDR/RR-TB is maintained with the BPaLM regimen (for 26 weeks).
  The dosage of each medication is as follows:
  * Bedaquiline 400mg/day for the 2 weeks, 200mg/TIW afterward
  * Pretomanid 200mg/day
  * Linezolid 600mg/day for the 9weeks, 300mg/day afterward
  * Moxifloxacin 400mg/day

SUMMARY:
The objective of this study is to analyze the efficacy of a new regimen using Bedaquiline, Pretomanid, Linezolid, and Moxifloxacin for 24 weeks or Bedaquiline, Pretomanid, Linezolid for 26 weeks for the treatment of MDR/RR-TB through the clinical trial.

DETAILED DESCRIPTION:
The BPaL (Bedaquiline, Pretomanid, Linezolid) regimen has been proven effective for the treatment of Fluoroquinolone-resistant MDR-TB through studies such as the NixTB and ZeNix trials. In addition, the BPaLM regimen has been demonstrated to have excellent efficacy in RR-TB patients through the TB-PRACTECAL study. This study aims to analyze the efficacy of the BPaL(M) regimen in Korean MDR/RR-TB patients.

ELIGIBILITY:
Inclusion Criteria:

1. At least 19 years old at enrolment
2. Bodyweight over 35Kg
3. If rifampicin resistance is confirmed through molecular or phenotypic drug susceptibility testing conducted on sputum or bronchoscopy specimens within 3 months of screening
4. Chest radiological findings consistent with pulmonary tuberculosis

Exclusion Criteria:

1. Uncontrolled DM
2. Extrapulmonary TB that would require treatment longer than would be usual for pulmonary TB
3. Less than 30 Karnofsky score at enrolment
4. BMI less than 17
5. Known severe allergy to any of the BPaLM regimen drugs
6. Medical history of Glucose-galactose malabsorption, galactose intolerance, and Lapp lactase deficiency
7. HIV-positive
8. The QTcF interval exceeds 450 msec on the electrocardiogram at baseline
9. Patients who are at risk of Torsade de Pointes due to underlying heart diseases such as heart failure or arrhythmia
10. For women of childbearing potential if the pregnancy test is positive, women who are breastfeeding or planning to become pregnant within 6 months of discontinuation/termination of treatment during the study, or who do not want contraception (i.e., oral and subcutaneous hormonal contraceptives, condoms, diaphragms, intrauterine device, or use of appropriate contraceptive methods including abstinence)

    *Note: Double contraception (e.g., when a male uses a barrier contraceptive method such as a condom, a female partner uses a hormonal contraceptive or an additional contraceptive method such as an intrauterine device) is required while taking the study drug and up to 6 months after stopping/terminating the study drug. In particular, taking the study drug may affect the efficacy of hormonal contraceptives, and even if you are using only barrier contraception at the same time with your partner, you cannot be sure of preventing pregnancy, so it is necessary to maintain double contraception.
11. Men who plan to become pregnant during the study period or within 6 months of discontinuation/termination of treatment, or who do not wish to use double contraception or abstinence during this period.
12. Patients who have Grade 3 or 4 or higher peripheral neuritis, or Grade 1 or 2 with a high probability of progression to peripheral neuritis,
13. Current use of monoamine oxidase Inhibitor or used 2 weeks before treatment
14. Use of serotonergic antidepressant within 3 days of treatment
15. Any contraindication that may affect QTc interval (amiodarone, chloroquine, chlorpromazine, clarithromycin, haloperidol, etc.)
16. Any contraindication that may cause myelosuppression
17. Taking drugs that affect the cytochrome P450 enzyme within 30 days (quinidine, tyramine, ketoconazole, fluconazole, testosterone, quinine, gestodene, metyrapone, phenelzine, doxorubicin, troleandomycin, cyclobenzaprine, erythromycin, cocaine, furafylline, cimetidine, dextromethorphan, etc.)
18. Previously treated with Bedaquiline or Linezolid for more than 4 weeks
19. Abnormal value of a blood test at baseline:

    * Hypokalemia, Hemoglobin < 8.0 g/dL, Platelet < 75,000/mm3, ANC < 1000/mm3
    * AST or ALT > 3 X ULN, Total bilirubin >2.0 X ULN, Albumin < 3.2 mg/dL
    * Serum creatinine > 2 X ULN, Serum calcium < LLN, Serum magnesium < LLN

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-12-13 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
A microbiological failure or clinical failure or relapse | until 12 months after the end of treatment
  A microbiological failure or clinical failure or relapse during the treatment period and the 12-month follow-up period after end of treatment

SECONDARY OUTCOMES:
Time to sputum culture conversion during the treatment period | 26 weeks or 24 weeks
  Analyze the time to liquid and solid culture conversion and estimate the median value using the Kaplan-Meier Method
Proportion of culture-negative patients at specific times (weeks 4, 8, 12, 16, and 24 or 26) | 26 weeks or 24 weeks
  Frequency analysis of liquid and solid culture conversion at a specific time point
Prescribed dose of Linezolid | 26 weeks or 24 weeks
  Analyze the actual dose of linezolid prescribed
All-cause mortality | 26 weeks or 24 weeks
  Analyze the frequency and fraction of deaths and estimate the median using the Kaplan-Meier Method

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, Songpa-gu, South Korea

IPD SHARING:
Plan to Share IPD: No